CLINICAL TRIAL: NCT02987036
Title: Administration of Beta-agonistic Drug Using Two Different Nebulizer Technologies: Effects on Lung Mechanics
Brief Title: Delivery of Beta Agonists is Technique Sensitive (DOBATS)Mechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Dr., Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: nebulizer
Record Dates: First submitted 2016-01-13; First posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Respiratory Failure
Keywords: nebulizer technologies, lung mechanics, beta-agonistic drug
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerogen (Experimental): Two doses of aerosolized Albuterol sulfate (2.5 mg dissolved in saline) At study start (T l 0) and after 6 hours (Tll0) by Aerogen
  Interventions: Device: Aerogen
- Jet Nebulizer (Other): Two doses of aerosolized Albuterol sulfate (2.5 mg dissolved in saline) At study start (T l 0) and after 6 hours (Tll0) by Jet Nebulizer
  Interventions: Device: Jet nebulizer

INTERVENTIONS:
Device: Aerogen — Two doses of aerosolized Albuterol sulfate (2.5 mg dissolved in saline) At study start (T l 0) and after 6 hours (Tll0) by mesh nebulizer
  Arms: Aerogen
Device: Jet nebulizer — Two doses of aerosolized Albuterol sulfate (2.5 mg dissolved in saline) At study start (T l 0) and after 6 hours (Tll0) by Jet nebulizer
  Arms: Jet Nebulizer

SUMMARY:
The purpose of this study is to find out weather differences in administration nebulizer technology (Jet nebulizer VS. mesh nebulizer) will have impact on lung mechanic variables (Compliance, resistance and PEEPi) during controlled mechanical ventilation.

DETAILED DESCRIPTION:
The delivery of aerosols has a two fold appeal as it is distributed direct to the tracheo- bronchial tree and alveolar epithelium. The drug is then rapidly absorbed by the circulation avoiding the first pass entero-hepatic metabolic effect.

The systemic effects may be regarded as a side effect in the case were the primary therapeutic target is aimed at the bronchial tree as is the case with broncho-active drugs, such as β2-stimulants.

The ability of particles to remain suspended in a gas can be predicted from their size, shape and density, coupled with the density and viscosity of the gas. The properties of an aerosol is commonly expressed as the Mass Median Aerosol Diameter MMAD, a measure of the average particle size and the geometric standard deviation. It is calculated from the cumulative particle size curve1. The MMAD will give a reliable estimate of the likely deposition of the drug along the tracheo-bronchial tree. A particle size >5 will likely deposit in the upper airways, while particles with an MMAD of 2-5 is likely to deposit in the tracheo-bronchial tree2.

Jet nebulizers are the most commonly used devices for aerosol therapy. However, the MMAD generated by this device is unpredictable, often leading to the drug being deposited in the ventilator circuit or endotracheal tube3.

An alternative is the vibrating mesh nebulizer, which is based on a high frequency vibrating piezoelectric crystal. The crystal will vibrate a micron mesh at a very high frequency. A micro pump will deliver a small volume of liquid from a reservoir into the vibrating mesh resulting in a very precise aerosol generation3.

Nebulizer therapy is often prescribed without proven effects or proper evaluation of result. Indeed, two large multicenter trial in acute lung injury patients were discontinued at interim analyses due to lack of effect4,5. This lack of effect may be due to the nebulizer technology (Jet nebulizer), the indication (ARDS), or primary outcome.

The investigators would like to compare the difference in therapeutic effect between these two devices as this has not been published previously. It is well known that the physical properties of the generated aerosol may differ widely, depending on device and technology used. Hence, even if the same amount of drug is administered, distribution and uptake will not be the same. It can further be expected that the therapeutic response will be different.

ELIGIBILITY:
Inclusion Criteria:

* Patients on mechanical ventilation for more than 48 hours
* PEEPi ≥3 cm H2O and expected to remain on controlled mechanical ventilation for at least 24 hours.

Exclusion Criteria:

* Severe chronic lung disease with chronic hypercapnia (PCO2>45 mm Hg), Chronic hypoxemia (PO2< 55mm Hg with FiO2=0,21), hospitalization within last 6 months for respiratory failure (PCO2>50; PO2<55mm Hg), Secondary polycythemia, severe pulmonary hypertension (mPAP >40 mm Hg.
* Unable to obtain consent
* Acute myocardial infarction
* Severe congestive heart failure
* Heart rate greater than maximal predicted heart rate MHR85 (MHR 85=0.85 x (220-age).
* Burns over more than 40% of body surface area
* Cancer or other irreversible disease or condition for which 6-month mortality is estimated to be greater than 50%
* Allogenic bone marrow transplantation within 5 years prior to the study
* Diffuse alveolar hemorrhage from vaculitis
* Morbid obesity
* Moribund, not expected to survive 24 hours
* Daily use of beta agonists prior to hospitalization
* Participation in other study
* Chronic liver disease
* Neuromuscular disease that impairs ability to breath without assistance (e.g. Cervical spine cord injury at level C5 and higher, Amyotrophic lateral sclerosis, Guillain-Barre syndrome or myasthenia gravis)
* Pregnant or breast-feeding

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
change of intrinsi PPPE | 0, 5min, 60min, 6h after the first administration; 5min, 60 min and 18 h after second administration

SECONDARY OUTCOMES:
change of respioratory resistance | 0, 5min, 60min, 6h after the first administration; 5min, 60 min and 18 h after second administration
change of respiratory system Compliance | 0, 5min, 60min, 6h after the first administration; 5min, 60 min and 18 h after second administration

CONTACTS AND LOCATIONS:
Overall Officials: Ling Ling, Dr, Study Director — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No